CLINICAL TRIAL: NCT00891514
Title: Aging, Inflammation and Exercise in Chronic Stroke
Brief Title: Trial of Aerobic Exercise Training in Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alice S. Ryan, PhD, Professor, Baltimore VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0118; R01AG030075 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Stroke; Insulin Resistance; Sedentary Lifestyle
Keywords: Exercise; Inflammation; Insulin Sensitivity
MeSH Terms: conditions — Stroke; Insulin Resistance; Sedentary Behavior; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (Experimental): Treadmill training
  Interventions: Behavioral: Aerobic Exercise
- Stretch Control (Active Comparator): Stretching exercises
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Aerobic Exercise — Treadmill training- begins at 15 minutes total duration at 40-50% maximal heart rate reserve 3 times per week, increasing to 60-70% maximal heart rate reserve for 45-60 minutes for 6 months
  Arms: Aerobic Exercise
Behavioral: Stretching — Stretching, balance exercises, and components of conventional physical therapy-- begins at 15 minutes and progresses to 45 minutes for 6 months
  Arms: Stretch Control

SUMMARY:
The purpose of this study is to examine the effects of treadmill training on inflammation in the skeletal muscle and adipose tissue, insulin action in the skeletal muscle, and whole body glucose metabolism in stroke survivors. The fundamental hypothesis of this study is that key inflammatory markers in adipose tissue and skeletal muscle are abnormal, skeletal muscle insulin signaling is impaired, and systemic insulin sensitivity is reduced in hemiparetic stroke patients and that these factors are modifiable and improved by exercise training in stroke patients.

DETAILED DESCRIPTION:
Many stroke survivors are sedentary and are at risk for the development of diabetes. We will study the interactions of adipose tissue and the paretic and non-paretic muscle inflammation, insulin signaling and action in hemiparetic stroke patients and the ability to employ exercise training to reverse these abnormalities in this ethnically diverse population. Participants aged 40-75 years with chronic stroke will be randomized to treadmill training versus stretch control group using a one-two-one blocked randomization on race (black vs. white), sex (male vs. female), and glucose tolerance status (normal vs. impaired and type 2 diabetes).

Stroke occurs in over 780,000 persons each year in the U.S., the vast majority reported in persons older than 55 years of age. Following stroke, patients remain at continued high risk for recurrent stroke. Inflammatory processes lead to cardiovascular events/stroke and contribute to disease risk progression by impacting insulin resistance and the development of type 2 diabetes. Interventions that reduce inflammation and improve insulin sensitivity have important clinical implications, especially in the stroke population.

Task-oriented treadmill training is utilized to improve cardiovascular fitness and functional mobility in hemiparetic stroke patients. Additionally, preliminary data indicates that progressive treadmill training in this population improves glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke greater than or equal to 6 months prior with stable residual hemiparetic gait deficits
* Already completed all conventional inpatient and outpatient physical therapy
* Adequate language and neurocognitive function to safely participate in exercise testing and training
* Men or women ages 40-75 years
* Body mass index between 20 to 50 kg/m2
* Non-smoker, or history of no smoking for more than 5 years
* Under the care of a primary care medical provider

Exclusion Criteria:

* Already performing aerobic exercise 3 times a week
* Increased alcohol consumption defined as greater than 2 oz. liquor or 8 oz. of wine or 24 oz. of beer per day
* Cardiac history of:

  1. unstable angina
  2. recent (less than 3 months prior to study entry) myocardial infarction, congestive heart failure
  3. hemodynamically significant valvular dysfunction
* Medical History:

  1. recent hospitalization (less than 3 months prior to study entry) for severe medical disease
  2. peripheral arterial disease with vascular claudication
  3. orthopedic or chronic pain condition restricting exercise
  4. pulmonary or renal failure
  5. active cancer
  6. untreated poorly controlled hypertension measured on at least 2 occasions (greater than 160/100)
  7. type I diabetes mellitus, insulin therapy, untreated and/or poorly controlled diabetes with fasting blood glucose of greater than 160
  8. smoking within the last 5 years
  9. allergy to lidocaine
  10. medications: heparin, warfarin, lovenox, beta-blockers, oral steroids
* Neurological history of:

  1. dementia with Mini-Mental Status Score less than 23 (less than 17 if education level at or below 8th grade), and diagnostic confirmation by neurologist or psychiatrist
  2. severe receptive or global aphasia which confounds testing and training, operationally defined as unable to follow 2 point commands
  3. hemiparetic gait from a prior stroke preceding the index stroke defining eligibility (more than one stroke)
  4. neurologic disorder restricting exercise, such as Parkinsons Syndrome or myopathy
  5. untreated major depression
* Adipose tissue and muscle biopsy exclusion criteria:

  1. anti-coagulation therapy with heparin, warfarin, or lovenox (anti-platelet therapy is permitted)
  2. bleeding disorder
  3. allergy to lidocaine

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
VO2peak | Baseline and 6 months
  maximal oxygen consumption during a treadmill test

SECONDARY OUTCOMES:
Whole body insulin sensitivity | Baseline and 6 months
  glucose utilization during a glucose clamp
Cytokines | Baseline and 6 months
  circulating TNF alpha levels
Body fat | Baseline and 6 months
  whole body percent fat
Muscle mass | Baseline and 6 months
  whole body lean mass

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — University of Maryland, VA Research Service; Charlene Hafer-Macko, MD, Principal Investigator — University of Maryland, VA Research Service, Department of Neurology
Locations (1):
- University of Maryland, VAMC, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ryan AS, Dobrovolny CL, Smith GV, Silver KH, Macko RF. Hemiparetic muscle atrophy and increased intramuscular fat in stroke patients. Arch Phys Med Rehabil. 2002 Dec;83(12):1703-7. doi: 10.1053/apmr.2002.36399. PMID 12474173
- [Background] Hafer-Macko CE, Yu S, Ryan AS, Ivey FM, Macko RF. Elevated tumor necrosis factor-alpha in skeletal muscle after stroke. Stroke. 2005 Sep;36(9):2021-3. doi: 10.1161/01.STR.0000177878.33559.fe. Epub 2005 Aug 18. PMID 16109906
- [Background] Ivey FM, Ryan AS, Hafer-Macko CE, Goldberg AP, Macko RF. Treadmill aerobic training improves glucose tolerance and indices of insulin sensitivity in disabled stroke survivors: a preliminary report. Stroke. 2007 Oct;38(10):2752-8. doi: 10.1161/STROKEAHA.107.490391. Epub 2007 Aug 16. PMID 17702957
- [Derived] Ryan AS, Novitskaya M, Treuth AL. Predictive Equations Overestimate Resting Metabolic Rate in Survivors of Chronic Stroke. Arch Phys Med Rehabil. 2022 Jul;103(7):1352-1359. doi: 10.1016/j.apmr.2022.01.155. Epub 2022 Feb 19. PMID 35192798
- [Derived] Serra MC, Balraj E, DiSanzo BL, Ivey FM, Hafer-Macko CE, Treuth MS, Ryan AS. Validating accelerometry as a measure of physical activity and energy expenditure in chronic stroke. Top Stroke Rehabil. 2017 Jan;24(1):18-23. doi: 10.1080/10749357.2016.1183866. Epub 2016 Jun 20. PMID 27322733